CLINICAL TRIAL: NCT00011284
Title: Mechanisms of Inflammatory Liver Injury
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Other Study IDs: 6091-CP-001
Record Dates: First submitted 2001-02-15; First posted 2001-02-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2002-09

CONDITIONS: Liver Diseases
Keywords: Liver; Inflammation; Endotoxin; Neutrophils; Hepatocytes
MeSH Terms: conditions — Liver Diseases; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other

SUMMARY:
White blood cells can cause liver damage if they inappropriately accumulate in the liver in large numbers. Such an event can occur if an individual's blood is exposed to endotoxin, a substance released from the cell walls of many species of bacteria. The purpose of this study is to isolate neutrophils, an important white blood cell, from the blood of normal volunteers, and put them in tissue culture with isolated liver cells. The experiments will determine how endotoxin can increase the ability of neutrophils to damage liver cells. All studies supported by this grant will be done with isolated cells in tissue culture. This experimental model will reveal possible mechanisms that can in the future be evaluated in human diseases such as bacterial sepsis.

DETAILED DESCRIPTION:
Neutrophils will be isolated from normal human volunteers and placed in cell culture with isolated hepatocytes or C3A cells (hepatoblastoma cell line that exhibit many characteristics of normal hepatocytes). These experiments will evaluate the mechanisms by which neutrophil adhere to the surface of hepatocytes, and the mechanisms by which the attached neutrophils can damage or kill the hepatocytes. Mechanisms of adhesion will involve understanding of the chemokines released by the hepatocytes that stimulate neutrophil adhesiveness, the cytokines that activate hepatocytes to express chemokines and adhesion molecules, the adhesion receptors on the neutrophil surface that are able to recognize the adhesion molecules on the hepatocyte surface, and the ability of adhesion to enhance and focus cytotoxic chemicals coming from the stimulated neutrophils. In addition, the role endotoxin can play in these sequence of events is being studies, and the specific cytotoxic mechanisms released by the neutrophils are under study. As noted in the brief summary, this grant only supports use of human cells in vitro (i.e., all experiments will be done in tissue culture). The purpose of working with this experimental model is to define what mechanisms should in future experiments be evaluated in patients with endotoxin induced disease.

ELIGIBILITY:
Only blood from normal subjects will be used in the in vitro experiments.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Study Completion 2001-11

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States